CLINICAL TRIAL: NCT06272760
Title: Development and Validation of a Remote Therapy Protocol Using Multimodal Sensor Fusion for Upper Limb Function Enhancement in Children With Cerebral Palsy
Brief Title: Development of a Remote Therapy Protocol for Upper Limb Function Enhancement in Children With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeong Yi Kwon, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-02-060
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Physical activity; Telerehabilitation; Accelerometer
MeSH Terms: conditions — Cerebral Palsy; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Single blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tele-HABIT (Experimental): Children in the experimental group are going to receive intensive bimanual activity-based occupational therapy, known as Home-Based HABIT (H-HABIT). This therapy is going to be administered remotely. Each session will last for 2 hours and was conducted 5 times a week. The total duration of this intervention is 3 weeks.
  Interventions: Other: Home-based hand-arm bimanual intensive training (Tele-HABIT)
- Control (No Intervention): Children in the control group will not receive any intervention during the 3-week study period. They will be placed on a waitlist and offered the same therapy after the study is completed.

INTERVENTIONS:
Other: Home-based hand-arm bimanual intensive training (Tele-HABIT) — Hand-Arm Bimanual Intensive Therapy (HABIT) is a therapeutic approach designed to improve the motor skills and functional use of both arms in individuals with conditions such as cerebral palsy. The core principle of HABIT is to encourage voluntary exercise by actively engaging the affected side, which may be weaker or partially paralyzed, in various activities. This approach aims to reduce physical and mental discomfort while maximizing the effectiveness of the training. HABIT has been adapted into a home-based format by ZOOM, referred to as Home-Based HABIT (H-HABIT).
  Arms: Tele-HABIT

SUMMARY:
The perpose of this study: Development and demonstration of a teletherapy protocol to improve upper limb function in children with cerebral palsy.

DETAILED DESCRIPTION:
* Development of a home-based remote upper limb function evaluation program using heterogeneous (multimodal) sensors.
* Development of a home-based remote upper limb function improvement treatment program using heterogeneous sensors.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 12 years
* MACS level 1-4
* Diagnosed with CP due to central nervous system lesions

Exclusion Criteria:

* Individuals with a Manual Ability Classification System (MACS) level V, indicating an inability to use both hands in daily life activities.
* Individuals who fall within levels 0 to 4 of the House Functional Classification System.
* Individuals with severe intellectual disabilities, characterized by difficulties in understanding or following instructions.
* Individuals with vision impairment that could affect participation in the therapy.
* Individuals who have received a botulinum toxin injection in the upper extremity within the past 6 months.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from Assisting Hand Assessment (AHA) score at post-intervention test (T1-T0). | Baseline and 1 month (post intervention)
  AHA is a standardized tool for children(18 months-12 years) with unilateral CP. The AHA measures the child's ability to use the affected hand to assist the unaffected hand in a variety of bimanual activities. The 15-20 minute session uses semi-structured play with specific items. A certified AHA assessor views the videorecording to score the child's displayed willingness and ability to use the weaker arm and hand on each of 22 items from 1 (= does not do) to 4 (= effective). The AHA has inter- and intra-rater reliabilities of 0.98 and 0.97 respectively and content validity established during initial development. For data analysis, we generated AHA Logit scores (as recommended in the administration manual) that transform the raw (ordinal) scores into interval level data.

SECONDARY OUTCOMES:
Change from Baseline Pediatric Motor Activity Log (PMAL) score at post-intervention test (T1-T0). | Baseline and 1 month (post intervention)
  The PMAL was derived from the Motor Activity Log, which is used as an assessment tool in adults who participated CIMT, to measure changes in upper extremity use in real life. This parental assessment tool rates the use of the children's affected upper extremities in daily activities. Twenty-two arm-hand functional tasks that are typical for children aged 7 months to 8 years (e.g., taking off socks or shoes, holding a cup) were assessed and collected as a systemic data. The test has two components: (1) how often (PMAL HO) and (2) how well (PMAL HW). Parents rate PMAL HO on a 6-point scale from 0 (not at all) to 5 (all the time) and PMAL HW from 0 (does not use) to 5 (same as the unaffected arm). This tool has a high test-retest reliability (r=0.94; P<0.01) and a high internal consistency (Cronbach's α=0.88 to 0.95).
Change from Baseline Melbourne Assessment 2 (MA2) score at post-intervention test (T1-T0). | Baseline and 1 month (post intervention)
  The Melbourne Assessment 2 (MA2) is a specific upper limb assessment focusing on the capacity of one hand. It benchmarks against certain criteria, delving into facets like movement range, accuracy, agility, and flow. The test was videotaped for analysis, and the raw score converted to a percentage of the maximal score.The higher the score, the better the motor function is interpreted. Test-retest results revealed moderate to high intrarater reliability for item totals (mean of 0.83 and 0.79) for each rater and high reliability for test totals (0.98 and 0.97).
Change from Canadian Occupational Performance Measure (COPM) score at post-intervention test (T1-T0). | Baseline and 1 month (post intervention)
  The COPM was designed as an outcome measure with a semi-structured interview format and structured scoring method to assess a person's level of self-efficacy. It conceptualizes self-efficacy in terms of self-perception of performance and satisfaction with performance. The COPM uses three 10-point rating scales to rate importance, performance and satisfaction. A score value of '1' refers to a low rating (i.e. 'not important at all', not able to do it at all', 'not satisfied at all'). A score value of '10' refers to a high rating (i.e. 'extremely important', 'able to do it extremely well', 'extremely satisfied'). Summing the ratings across problems and dividing by the total number of problems derive separate total performance and satisfaction scores.
Change from Pediatric Evaluation of Disability Inventory Computer Adaptive Test (PEDI-CAT) score at post-intervention test (T1-T0). | Baseline and 1 month (post intervention)
  The Pediatric Evaluation of Disability Inventory Computer Adaptive Test (PEDI-CAT) was developed to respond to the need for an accurate and efficient functional measure with content for children and youth in multiple functional content areas. The new PEDI-CAT measures function in the three domains of Daily Activities, Mobility and Social/Cognitive for infants, children and youth from birth through 20 years of age. In addition, the PEDI-CAT's Responsibility domain measures the extent to which the caregiver or child takes responsibility for managing complex, multi-step life tasks. The higher the score, the better the functional ability is interpreted.
Change from baseline Magnitude ratio (Accelerometer) at post-intervention test (T1-T0). | Baseline and 1 month (post intervention)
  The magnitude ratio is calculated as a metric to compare the magnitude of acceleration of the arms at each time point: ln(paretic magnitude/nonparetic magnitude). The magnitude will be calculated by taking the vector magnitude of the activity counts for each epoch. The natural log will be used to avoid skewness in the ratio caused by an underestimation of the denominator. The average magnitude will be calculated for each period. A magnitude ratio near 0 indicates similar use of each arm, a negative number indicates more use of the nonparetic arm, and a positive number indicates more use of the paretic arm.
Change from baseline Bilateral magnitude(Accelerometer) at post-intervention test (T1-T0). | Baseline and 1 month (post intervention)
  The bilateral magnitude is used to compare the overall movement of both arms together as a measure of bilateral arm movement: nonparetic magnitude + paretic magnitude. As with the magnitude ratio, the vector magnitude of the activity counts will be calculated for each epoch. A greater bilateral magnitude indicates greater overall movement of both arms.
Quantitative Analysis of Ocular Motor Function Using a Wearable Eye-Tracking Device (Neon) | Baseline and 1 month (post intervention)
  This outcome assesses ocular motor function through the use of a wearable eye-tracking device (Neon; Pupil Labs GmbH, Germany). The Neon system records real-time eye movement parameters during standardized visual-perceptual and motor tasks without requiring calibration. Key variables include fixation duration, saccadic amplitude, pupil dilation, and gaze stability. Data will be used to identify oculomotor biomarkers that reflect potential deficits in visual-motor integration and central visual-vestibular processing in children with unilateral cerebral palsy. Eye-tracking recordings are synchronized with task performance and analyzed using validated software (Pupil Cloud). This objective measure is intended to complement clinical test scores and provide deeper insight into underlying sensorimotor integration difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: JEONG-YI KWON, MD, PHD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea